CLINICAL TRIAL: NCT03334565
Title: Reducing Particulate Matter-associated Cardiovascular Health Effects for Seniors
Brief Title: Reducing PM-associated CV Health Effects for Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Masako Morishita, Associate Professor, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R01NR014484 (NIH)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Diseases in Old Age

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham (Sham Comparator): Participants were exposed to unfiltered ambient air (sham) filtered air using air filtration systems in the bedroom and main living space of each residence.
  Interventions: Device: Air filtration systems without filters (sham)
- Low efficiency (Active Comparator): Participants were exposed to low-efficiency (LE) "HEPA-type" filtered air using air filtration systems in the bedroom and main living space of each residence.
  Interventions: Device: Low efficiency air filtration systems
- High efficiency (Active Comparator): Participants were exposed to high-efficiency (HE) "true-HEPA" filtered air using air filtration systems in the bedroom and main living space of each residence.
  Interventions: Device: High efficiency air filtration systems

INTERVENTIONS:
Device: Low efficiency air filtration systems — Subjects were exposed to low-efficiency filtered air.
  Arms: Low efficiency
Device: High efficiency air filtration systems — Subjects were exposed to high-efficiency filtered air.
  Arms: High efficiency
Device: Air filtration systems without filters (sham) — Subjects were exposed to unfiltered air.
  Arms: Sham

SUMMARY:
The objective of this study is to investigate the effectiveness of air filtration at reducing personal-level exposures to fine particulate matter (PM2.5) and mitigating related cardiovascular (CV) health effects among older adults in a residential facility in a representative US urban location.

We enrolled 40 nonsmoking older adults into a randomized double-blind crossover intervention study with daily CV health outcomes and PM2.5 exposure measurements. The study was conducted in a low-income senior living apartment building in downtown Detroit, Michigan.

Participants were exposed to three 3-day scenarios separated by one-week washout periods: unfiltered ambient air (control), low-efficiency (LE) "HEPA-type", and high-efficiency (HE) "true-HEPA" filtered air using air filtration systems in the bedroom and main living space of each residence.

The primary outcome was brachial blood pressure (BP). Secondary outcomes included noninvasive aortic hemodynamics and pulse wave velocity and heart rate variability. PM2.5 exposures were measured in the participants' residences as well as by personal-level monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 85 years old
* non-smoking healthy adults

Exclusion Criteria:

* smoke or anyone in your residence smokes.
* had a cardiovascular event within the past 6 months (such as myocardial infarction (heart attack), angina, cardiac or carotid surgery or stent, diagnosed peripheral arterial disease, aortic aneurysms, treated heart failure, any treated arrhythmia including atrial fibrillation)
* have renal disease requiring dialysis.
* have had medication changes in the past 6 weeks.
* use supplementary oxygen.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
brachial blood pressure | at the same time between 8-10 AM on 3 consecutive days starting 24 hours after filter system placement
  Brachial blood pressure was measured using a BPTru device.

SECONDARY OUTCOMES:
noninvasive aortic hemodynamics | at the same time between 8-10 AM on 3 consecutive days starting 24 hours after filter system placement
  Aortic hemodynamics was measured using a SphygmoCor device.
Pulse wave velocity | at the same time between 8-10 AM on 3 consecutive days starting 24 hours after filter system placement
  Pulse wave velocity was measured using a SphygmoCor device.
heart rate variability | at the same time between 8-10 AM on 3 consecutive days starting 24 hours after filter system placement
  Heart rate variability was measured using a SphygmoCor device.
microvasculature tone | at the same time between 8-10 AM on 3 consecutive days starting 24 hours after filter system placement
  Retinal photography was used to measure retinal arteriole diameters.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morishita M, Adar SD, D'Souza J, Ziemba RA, Bard RL, Spino C, Brook RD. Effect of Portable Air Filtration Systems on Personal Exposure to Fine Particulate Matter and Blood Pressure Among Residents in a Low-Income Senior Facility: A Randomized Clinical Trial. JAMA Intern Med. 2018 Oct 1;178(10):1350-1357. doi: 10.1001/jamainternmed.2018.3308. PMID 30208394